CLINICAL TRIAL: NCT00582218
Title: Family Access to Care Study (FACS)
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Bruce Rapkin, PhD, Memorial Sloan-Kettering Cancer Center
Other Study IDs: 03-008
Record Dates: First submitted 2007-12-21; First posted 2007-12-28 (Estimated); Last update posted 2009-01-14 (Estimated); Status verified 2009-01

CONDITIONS: HIV Infections
Keywords: HIV/AIDS; Access to care
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

SUMMARY:
The purpose of this study is to find ways to get services to families living with HIV. New services for families living with HIV have been tried in places around the country. They seem to benefit many families. We will work with places in New York City that provide HIV services to find out more about family services. There, we will talk with people living with HIV, their family members, and their providers. Many questions need to be answered. For example: What kinds of services do families want? What would make it easier for families to come in for services? What would get in the way?

DETAILED DESCRIPTION:
Families affected by HIV and AIDS require access to a comprehensive continuum of services. Findings from our own and other recently completed federally sponsored intervention trials and other studies could be used to help expand and enhance these services. However, a number of fundamental questions must first be answered about the feasibility of "technology transfer." This study will address this issue by conducting individual interviews and focus groups with providers from 64 medical care and social service settings. Data will also be obtained through a comprehensive assessment of providers' capacities to serve families and to participate in technology transfer, including dimensions of organizational mission and leadership, availability of resources, and connections in the community. Thirty patients/clients served by each setting along with approximately twenty of their family members will also be individually interviewed to assess their needs for services, factors that affect their desire for family-oriented services, and their willingness to take part in psychosocial intervention studies. Data analysis will determine how initial setting readiness and setting capacities, and feedback about patient and family needs and willingness to participate in research, influence change in readiness, interest in capacity building and participation in research partnership activities. We will also conduct hierarchical data analyses to better understand how providers' readiness and capacities are related to clients'and families' service needs, barriers to participation, and willingness to participate in research. Study findings will guide efforts to implement family-oriented intervention research in frontline community service settings, and will help to establish a scientific framework for studying the process of technology transfer. Additionally, this project will lay the groundwork for sustained research collaboration with the network of community providers participating in this study to further explore ways to address the needs of families affected by HIV/AIDS.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria for Sampling AIDS Care Settings: Our goal in sampling is to identify and recruit the kinds of organizations that might ultimately be targets for Phase IV trials and other Memorial Sloan-Kettering Cancer Center dissemination efforts. For purposes of this research, we define an "AIDS Care Setting" as any setting which:

* Provides primary medical care, case management, day treatment, mental health or substance use treatment for people living with HIV/AIDS.
* Includes two or more full-time professional staff (e.g., social workers, nurses, clergy, physicians, or psychologists) with primary responsibility for an HIV/AIDS population.
* Has an active caseload of at least 50 people with HIV/AIDS.
* Has been in operation as an HIV/AIDS provider for at least two years.
* Has leadership and staff who are agreeable to participate in the work plan outlined in the Memorandum of Understanding (MOU).

Inclusion Criteria for Providers:

* Working as an administrator of HIV/AIDS care services, or a direct provider of services to HIV+ patients/clients.
* Working at the agency for at least 6 months.
* Working at the agency at least 20 hours a week.
* Able to converse in English or Spanish.
* Identified by agency leadership as staff who meet above criteria and can be approached, or want to volunteer to be interviewed.

Inclusion Criteria for Sampling Patients/Clients:

* Identified as HIV+ (according to identification by setting staff and/or by virtue of receiving services in a program exclusively designated for people infected with HIV/AIDS).
* Receiving services at an HIV/AIDS Care Setting sampled for this study, at the time of recruitment.
* Identified as a setting client for at least three months (in order to answer questions about the setting).
* Age 18 or older or emancipated minors over age 16.
* Able to converse in English or Spanish.
* Physically and mentally capable of providing informed consent, as determined by a trained interviewer.

Inclusion Criteria for Patients'/Clients' Family Members: In keeping with the definition of family as "networks of mutual commitment" adopted by the NIMH Family and AIDS Consortium, and in recognition of the diverse types of family situations of people affected by HIV/AIDS, we will include anyone designated as a "family member" by the index client/patient who meets our other inclusion criteria:

* Identified by index patient client as "one of the people in my family most likely to participate in programs with me" at the HIV/AIDS Care Setting sampled for this study.
* Age 18 or older or emancipated minors over age 16.
* Able to converse in English or Spanish.
* Physically and mentally capable of providing informed consent, as determined by a trained interviewer.

Exclusion Criteria:

Exclusion Criteria for AIDS Care Settings: Note that two or more AIDS Care Settings may exist within a single institution or agency. For example, hospitals may have separate programs for adult and pediatric HIV. A community AIDS service organization may have multiple distinct programs for different populations. Also, two settings may be closely coordinated. In order to ensure independence among settings, we will adopt the following exclusionary criteria:

* Only one AIDS Care Setting administered or governed by a given institution will be included in the study. If one setting from a particular institution agrees to participate, other settings from that institution will be ineligible.
* Multi-site programs or programs of a single agency that are working together in a coordinated fashion for purposes of this study will be treated as a single "AIDS Care Setting." If we discover that programs are affiliated, we will remove them from the list. In general, we will attempt to carry out this project at the site initially identified, although involvement of multiple sites may be necessary.

Exclusion Consideration for Providers: All providers who are identified by the agency leadership will be approached. However, a provider will not be able to participate if he/she has already participated in the study as a provider from another agency.

Exclusion Considerations for Patients and Families: All patients/clients of settings identified for this study and meeting above inclusion criteria are eligible. Patients/clients will be able to participate regardless of whether or not they nominate a family member to participate in the study with them.

Patients/clients will not be able to participate if they:

* Are not HIV+.
* Have been receiving services at the HIV/AIDS care setting for less than three months.
* Are under the age of 18, or are not emancipated minors.
* Are not able to converse in either English or Spanish.
* Are physically and mentally incapable of providing informed consent, as determined by a trained interviewer.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients/clients and their families at HIV/AIDS care centers
Sampling Method: Non-Probability Sample
Enrollment: 3200 (Estimated)
Dates: Start 2003-02; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Rapkin, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org